CLINICAL TRIAL: NCT00029809
Title: Chinese Exercise Modalities in Parkinson's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: R01AT000612-01 (NIH)
Record Dates: First submitted 2002-01-23; First posted 2002-01-24 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Parkinson Disease
Keywords: Parkinsons Disease; Chinese exercise
MeSH Terms: conditions — Parkinson Disease

INTERVENTIONS:
Behavioral: Chinese exercise modalities

SUMMARY:
This study will compare the effects of two Chinese and one Western exercise modalities on the signs and symptoms of Parkinson's disease.

DETAILED DESCRIPTION:
The long-term goal of this project is to study the effects of different exercise modalities on Parkinson's disease (PD). PD is a disorder whose primary disability stems from motor dysfunction including balance. Recent studies have shown that the risk of falling in the elderly can be reduced through the practice of the Chinese complementary and alternative medicine (CAM) such as T'ai Chi Chuan (TCC). This finding may be highly significant to PD. Although a recent report from Emory suggests PD patients can do well with aerobic (walk-run) exercise training (AET), it is still unclear whether the potential anti-Parkinsonian effect of such modalities is secondary to improved physical fitness (CRF), motor control or both. CAM interventions such as TCC may offer a unique opportunity to examine these fundamental questions.

In PD we hypothesize that exercise training will reduce primary and secondary disability and that some of these changes represent adaptive reprogramming of central motor pathways. We will conduct a controlled double-blind, 16-week dose-response study of exercise based on caloric expenditure and thus on the cardiorespiratory fitness effects of exercise (CRF). The treatments will be Qi Gong (minimal caloric expenditure), TCC (low expenditure), and walk-cycle AET (moderate expenditure).

We will examine exercise-induced change in motor control using quantitative measures of motor disability, including dynamic gait stability measures. We will also examine exercise effects on central and peripheral indices of Parkinsonian motor disability.

A caloric "dose-response" effect of exercise would suggest CRF is a major determinant of the anti-Parkinsonian effects of exercise. If the Chinese modalities are as effective or superior to AET however, this would suggest that other mechanisms such as change in central motor programming may be playing a role (e.g. relaxation effects, reinforcement of central motor programs?). A better understanding of exercise-induced neural plasticity and motor control would offer a significant, and heretofore unexploited rehabilitative potential in PD.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients with Parkinson's Disease, defined as a clinical state in which at least two of these four cardinal features are present- 1) slowness of movement, 2) tremor at rest, 3) muscular rigidity, 4) gait disturbance or posture imbalance.
* Ambulatory patients with Parkinson's Disease not exercising regularly more than 2x per week. Willing to be randomly assigned to 1 of the 3 exercise modalities: Tai Chi, Qi Gong and Aerobic exercise.

NOTE THAT PARTICIPATION IN THE STUDY REQUIRES BI-WEEKLY PARTICIPATION IN A 16-WEEK SUPERVISED EXERCISE PROGRAM PLUS RELATED EVALUATIONS AT EMORY. ACCORDINGLY, RECRUITMENT IS LIMITED TO LOCAL PATIENTS.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Overall Officials: Jorge L. Juncos, MD, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886